CLINICAL TRIAL: NCT02792179
Title: A Pilot Longitudinal Follow-Up Study of Tau Burden in The Brain of Subjects With Alzheimer's Disease Who Previously Participated in Study BP29409 Using [18F]RO6958948 Positron Emission Tomography
Brief Title: Evaluation of [18F]RO6958948 as Tracer for Positron Emission Tomography (PET) Imaging of Tau Burden in Alzheimer's Disease Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BP39126
Record Dates: First submitted 2016-06-02; First posted 2016-06-07 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

ARMS (1):
- [18F]RO6958948 (Experimental): Each participant will receive a single intravenous (IV) dose of [18F]RO6958948 and a single PET scan approximately 9-24 months after the baseline scan (in Study BP29409).
  Interventions: Drug: [18F]RO6958948

INTERVENTIONS:
Drug: [18F]RO6958948 — Radiolabeled low molecular weight compound, administered as single IV injection. The mass dose of [18F]RO6958948 injected will be less than or equal to (</=) 10 micrograms (µg), injection volume </=20 mL. Target injected activity for [18F]RO6958948 will be 370 megaBecquerel (MBq) (10 millicurie [mCi]).

SUMMARY:
This is a longitudinal, follow-up study in participants with Alzheimer's disease (AD) who previously participated in study BP29409 (NCT02187627). This study is designed to assess the longitudinal change of Tau pathology in the brain of participants with AD using the PET ligand [18F]RO6958948 and to assess the safety and tolerability of PET ligand.

ELIGIBILITY:
Inclusion Criteria:

* AD participants previously scanned with [18F]RO6958948 in Roche Study BP29409
* Agreement to use highly effective contraception measures
* Body mass index (BMI) between 18 and 32 Kilograms per square meter (kg/m^2)
* A study partner able to accompany the participant to all visits and answer questions about the participant
* In the opinion of investigator, based on the medical history and physical examination, can safely tolerate tracer administration and the scanning procedures
* Documented positive visual read (as per local procedures for florbetapir or similar procedures for other amyloid tracers) of an amyloid PET scan, which in the opinion of the principal investigator is consistent with a diagnosis of AD

Exclusion Criteria:

Exclusion Criteria for All Participants

* History or presence of any clinically relevant hematological, hepatic, respiratory, cardiovascular, renal, metabolic, endocrine, or central nervous system disease or other medical conditions that are not well controlled, may put the participant at risk, could interfere with the objectives of the study, or make the participant unsuitable for participation in the study for any other reason in the opinion of the principal investigator
* Clinically relevant pathological findings in physical examination, electrocardiogram, or laboratory values at the screening assessment that could impact participant safety
* Known history of clinically significant infectious disease including autoimmune deficiency syndrome (AIDS) or serological indication of acute/chronic hepatitis B or C or Human Immuno Virus infection
* Women of childbearing potential must not be pregnant, or nursing and serum human chorionic gonadotropin (HCG) must be negative at the time of Screening Visit 1, and urine HCG must be negative on all subsequent visits
* Loss or donation of more than 450 milliliters (mL) blood in the 4 months before screening or donation of plasma within 14 days of screening
* Unsuitable veins for repeated venipuncture
* History of drug or alcohol abuse or positive result from urine screen for drugs of abuse
* Have received an investigational medication within the last 3 months or 5 times the elimination half-life, whichever is longer, prior to enrollment Exclusion Criteria Related to Trial Procedures
* Has had or is planning to have exposure to ionizing radiation that in combination with the study-related tracer administrations and scanning procedures would result in a cumulative exposure that exceeds the recommended annual exposure limit
* Presence of pacemakers; aneurysm clips; artificial heart valves; ear implants; foreign metal objects in the eyes, skin, or body, or any other circumstance that would contraindicate a magnetic resonance imaging (MRI) scan
* History of, or suffers from, claustrophobia or feels that he or she will be unable to lie still on their back in the MRI or PET scanner
* Has received treatment that targeted amyloid-beta or tau within the last 24 months

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-07-19 (Actual); Primary Completion 2016-09-28 (Actual); Study Completion 2016-09-28 (Actual)

PRIMARY OUTCOMES:
Regional Standardized Uptake Value (SUV), as Assessed by the tau PET Brain Scan | Day 1
Regional Standardized Uptake Value Ratios (SUVR), as Assessed by the Tau PET Brain Scan | Day 1
Change in SUV for Different Brain Regions | Baseline to approximately 24 months
Change in SUVR for Different Brain Regions | Baseline to approximately 24 months

SECONDARY OUTCOMES:
Percentage of Participants with Adverse Events | Screening to 7-14 days after Tau PET scan (Up to approximately 7 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Johns Hopkins Medical Institutions, Johns Hopkins Outpatient Center, Baltimore, Maryland, United States